CLINICAL TRIAL: NCT04202523
Title: Study of Combined Radiotherapy and Radiofrequency Ablation for Hepatocellular Carcinoma
Brief Title: Combined Radiotherapy and Radiofrequency Ablation for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangXiMU-HCC-RT&RFA
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation; Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT&RFA (Experimental)
  Interventions: Radiation: Radiofrequency ablation; Device: IMRT & SBRT
- RFA (Active Comparator)
  Interventions: Radiation: Radiofrequency ablation

INTERVENTIONS:
Radiation: Radiofrequency ablation — Liver cancer radiofrequency ablation is a clinical treatment method that uses electrode needles to penetrate the skin and liver into the tumor and completely destroy the tumor through the principle of heat production to achieve the purpose of treating tumors.
Device: IMRT & SBRT — Tumor radiation therapy is a local treatment method using radiation to treat tumors. Radiation includes alpha, beta, and gamma rays produced by radioactive isotopes and x-rays, electron beams, proton beams, and other particle beams produced by various types of x-ray therapy machines or accelerators. Current mainstream radiotherapy technologies include stereotactic radiation therapy (SRT). Stereotactic radiation therapy (SRT) includes three-dimensional conformal radiation therapy (3DCRT) and three-dimensional conformal intensity modulated radiation therapy (IMRT).
  Arms: RT&RFA

SUMMARY:
Liver cancer is a clinically high-grade malignant tumor, and the current incidence rate is increasing year by year. It has become the third most malignant tumor after gastric cancer and lung cancer, and has a high mortality rate. The patient's five-year survival rate is less than 8.5%, which the second leading cause of cancer death is a serious threat to the health of patients. Surgical resection is the preferred treatment plan for liver cancer. With the development of medical technology, the clinical efficacy of liver cancer has been significantly improved, but postoperative recurrence has not been effectively controlled. According to statistics, the recurrence rate of liver cancer after 5 years is as high as 77.0%. Even for small liver cancer resection, the recurrence rate is 40.0%~50.0% within 5 years after operation. At the same time, for recurrent liver cancer, surgical resection is still the preferred treatment plan, but affected by the location, size, distal metastasis and multi-center pathogenesis of liver cancer, only 10.4%~31.0% can be surgically removed. In recent years, RFA has been widely used in liver cancer and recurrent liver cancer due to its unique advantages such as minimally invasive, simple operation, wide indication, reproducible, low cost, and accepted by patients, and has achieved satisfactory results. However, study found that because of the special location of recurrent liver cancer, its multi-center origin, and the characteristics of intrahepatic micrometastasis, it is often accompanied by microvascular tumor thrombus (MVI), which greatly increases the risk of liver cancer recurrence. Moreover, since the treatment of RFA can only be effective for the local detection of recurrent foci, and the effect of detecting small lesions is poor, there is a higher risk of recurrence. The use of radiation therapy is getting more and more attention, and it is changing from the past palliative treatment to current curable treatment. From an oncologic point of view, a narrow margin <1 cm and microvascular invasion is not safe and is often associated with higher rates of recurrence and shorter patient survival. On the other hand, it is also believed that most intrahepatic recurrences arise from multicentric carcinogenesis and are distant from the resection margin.

Whether combined radiotherapy and RFA treatment of liver cancer and recurrent liver cancer can further improve the clinical efficacy, there are few reports. Therefore, the short-term and long-term effects of radiotherapy combined with RFA in the treatment of liver cancer and recurrent liver cancer are studied to provide guidance for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. According to the diagnosis and treatment of primary liver cancer (2017 version), patients diagnosed as primary liver cancer; 2, after surgery, CT or MRI and other related imaging examinations suggest recurrence of liver cancer and can not exclud micro lesions; 3. There is no history of systemic liver cancer chemotherapy and large vessel embolism; 4. Child-Pugh classification of liver function is grade A or B, and no xternal liver metastasisoccurs; 5, no serious cardiovascular or cerebrovascular diseases, renal or pulmonary organ disease; 6, no other malignant tumors; 7. all volunteered to participate in the study and signed informed consent.

Exclusion Criteria:

1, with hepatic encephalopathy, refractory ascites and other serious complications; 2, combined with serious blood system diseases; 3, pregnant or lactating women; 4, during the period of receiving other treatment measures; Those who refused follow-up or follow-up data were not confirmed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 2 years

SECONDARY OUTCOMES:
OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- TaoBai, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No